CLINICAL TRIAL: NCT03059784
Title: Mobile Application-based Multifaceted Management to Improve Long-term Care After Percutaneous Coronary Intervention
Brief Title: APP-based Multifaceted Management After PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yongjian Wu, Associate director of Coronary Artery Disease Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016-ZX16
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): APP-based multifaceted management, including sending education material, everyday medication reminder, giving risk factor control support, clinical support to patients after PCI through APP.
  Interventions: Other: APP-based multifaceted management
- control (No Intervention): usual care without APP

INTERVENTIONS:
Other: APP-based multifaceted management — Patients after PCI will be regularly given education materials, medication reminders, life-style behaviors instruction through APP. Cardiologists can interact with patients on advice provision and clinical support after discharge through APP.
  Arms: intervention

SUMMARY:
High rates of recurrent cardiovascular events and readmission after percutaneous coronary intervention (PCI) are important issues. Guidelines emphasize rehabilitation and secondary prevention. But many patients are lack of effective management after PCI.This study is aimed to examine the effect of mobile application (APP)-based multifaceted management on the improvement of long-term care after PCI.

DETAILED DESCRIPTION:
This is a cluster-randomized controlled trial to evaluate the effect of APP-based multifaceted management strategy on improvement of long-term care for medication adherence,risk factor control, and reduction of adverse events, readmission rate and mortality after PCI.It includes knowledge education, medication reminder,advice provision, support to change lifestyle behaviors. The program is interactive between care provider and patients. A total of 20 wards will be randomly assigned to intervention or usual care.Anticipated 1100 patients after PCI will be participated in the trial. All the participants will be followed up until 12 months.

ELIGIBILITY:
Inclusion Criteria:

* patients who have received percutaneous coronary intervention and are discharged alive in the study centers;
* patients who are able to use APP;
* patients who provide informed consent.

Exclusion Criteria:

* patients who are not able to use APP;
* dementia;
* mental disturbed;
* patients who are not willing to receive management and follow up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
evidence-based medication adherence (the proportion of participants taking 3 medications (aspirin, P2Y12 receptor inhibitor, statin) without contraindications) | at 12 months after PCI
  the proportion of participants taking 3 medications (aspirin, P2Y12 receptor inhibitor, statin) without contraindications

SECONDARY OUTCOMES:
rate of LDL-C achieving target | at 12 months after PCI
  rate of LDL-C achieving target based on guideline
rate of systolic blood pressure achieving target | at 12 months after PCI
  rate of systolic blood pressure achieving target based on guideline
readmission rate | 12 months after PCI
  readmission rate after PCI

OTHER OUTCOMES:
smoking status (the proportion of participants with smoking cessation) | at 12 months after PCI
  the proportion of participants with smoking cessation
rehabilitation (the proportion of participants who receive rehabilitation program) | 12 months after PCI
  the proportion of participants who receive rehabilitation program

CONTACTS AND LOCATIONS:
Overall Officials: Yongjian Wu, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital

IPD SHARING:
Plan to Share IPD: Yes
management methods,outcomes including medication use, events of patients can be available on request.

REFERENCES:
- [Background] 1. Levine GN, et al. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention. Circulation. 2011,124:e574-e651 2. Kolh P, et al. 2014 ESC/EACTS Guidelines on myocardial revascularization. EHJ. 2014,35:2541-2619 3. Chow CK, et al. Effect of Lifestyle-Focused Text Messaging on Risk Factor Modification in Patients With Coronary Heart Disease: A Randomized Clinical Trial. JAMA, 2015, 314:1255-1263 4. Tian M, et al. A Cluster-Randomized, Controlled Trial of a Simplified Multifaceted Management Program for Individuals at High Cardiovascular Risk (SimCard Trial) in Rural Tibet, China, and Haryana, India. Circulation. 2015;132:815-824